CLINICAL TRIAL: NCT06742567
Title: Apixaban Prophylaxis for Prevention of Left Ventricular Thrombus Following Anterior Myocardial Infarction: An Open Label, Randomized Clinical Trial (POTAMI)
Brief Title: Apixaban Prophylaxis for Prevention of Left Ventricular Thrombus Following Anterior Myocardial Infarction
Acronym: POTAMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Professor Abdul Hakeem, professor, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-83/2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Acute Myocardial Infarction of Anterior Wall; Left Ventricular Thrombus; Prophylaxis
Keywords: Acute myocardial infarction; severe left ventricular dysfunction; prevention of LV thrombus; DOAC; apixaban
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Ventricular Dysfunction, Left | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Eligible patients will be enrolled after informed consent. Randomization will be undertaken once post primary PCI echocardiography is done and LV function is recorded. Patients with anterior wall myocardial infarction with severe left ventricular dysfunction defined by an EF<35% without evidence of LV thrombus will be screened. Patients randomized to the treatment arm will be given Apixaban 2.5 mg twice daily and DAPT for two weeks in addition to other guideline directed medical therapy (GDMT). After two weeks of triple therapy (DOAC+DAPT), aspirin will be dropped in the study arm. The control arm will be standard DAPT and GDMT without apixiban.
  Primary endpoint will be the incidence of left ventricular thrombus in the study arm vs the control group at one month echocardiographic follow up. While an open label trial, end point adjudication will be blinded where the echocardiographer will not know treatment allocation of the two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Apixaban 2.5 mg bid) (Experimental): Patients randomized to the treatment arm will be given Apixaban 2.5 mg twice daily and DAPT (aspirin (75 mg) + clopidogrel (75 mg)) for four weeks in addition to other guideline directed medical therapy (GDMT). After 4 weeks, treatment group will be switched to DAPT. o In the event of stent thrombosis during the study period, considering the high ischemic risk, the patient will be switched to ticagrelor instead of clopidogrel, and aspirin will be discontinued while Apixaban will be continued. After four weeks, the patient will be switched to DAPT (aspirin
  + ticagrelor).
  Interventions: Drug: Apixaban 2.5 MG PO BID
- Control group (Active Comparator): The control arm will be of standard care i.e. DAPT in addition to other guideline directed medical therapy (GDMT).
  Interventions: Drug: Control (Standard treatment)

INTERVENTIONS:
Drug: Apixaban 2.5 MG PO BID — Patients randomized to the treatment arm will be given Apixaban 2.5 mg twice daily and DAPT (aspirin (75 mg) + clopidogrel (75 mg)) for four weeks in addition to other guideline directed medical therapy (GDMT). After 4 weeks, treatment group will be switched to DAPT.
  Arms: Study arm (Apixaban 2.5 mg bid)
Drug: Control (Standard treatment) — DAPT plus guideline directed medical therapy
  Arms: Control group

SUMMARY:
The objective of this randomized controlled trial is to compare the safety and efficacy of low dose Apixaban (2.5 mg bid) in addition to guideline directed medical therapy vs guideline directed medical therapy alone in the prevention of left ventricular thrombus formation (after 30-days) following primary PCI in patients with acute anterior myocardial infarction with severe LV dysfunction.

DETAILED DESCRIPTION:
Objective To compare the safety and efficacy of Apixaban vs. placebo in the prevention of LV thrombus formation in patients with acute anterior myocardial and severe LV dysfunction following primary PCI in an open label, randomized controlled trial.

Methods:

Inclusion Criteria .Patients aged 18-65 years, presenting with acute anterior STEMI and severe LV dysfunction (EF<35%) with antero-apical akinesis, dyskinesis, or aneurysm.

Exclusion Criteria

* Patients with previous myocardial infarction or revascularization procedures.
* Patients with cardiogenic shock
* Patients with advanced CKD (Cr < 2 and those on hemodialysis)
* Recent ICH or major bleed requiring transfusion, low platelet counts<100,000
* History of CVA
* Patients with atrial fibrillation or other indications for chronic anticoagulation
* Pregnant patients and those with hematological disorders

Eligible patients will be enrolled after informed consent. Randomization will be undertaken once post PCI echocardiography is done and LV function is recorded. Patients randomized to the treatment arm will be given Apixaban 2.5 mg twice daily and DAPT for two weeks in addition to other guideline directed medical therapy (GDMT). After two weeks of triple therapy (DOAC+DAPT), aspirin will be dropped in the study arm. The control arm will be of standard care. After 4 weeks, treatment group will be switched to DAPT.

Follow up The primary endpoint will be the incidence of LV thrombus formation recorded at 4-week follow-up echocardiography. Patients' clinical status, side effects, and medication compliance will be recorded.

At 2-week: patients will be contacted via phone call to assess their clinical status, ensure drug compliance, discuss any necessary changes in drug regimen for those in the treatment group already prescribed on discharge, and inquire about any side effects.

At 4-week: patients will undergo an in-person follow-up where echocardiography will be conducted alongside a comprehensive assessment In case of any cardiac complaints, patients will be advised to visit the hospital or cardiologist promptly to complete a comprehensive clinical and laboratory workup. Primary endpoint

. Incidence of LV thrombus formation in the treatment arm vs. placebo at 4 week follow up echocardiography.

Secondary endpoints

* composite of death, recurrent myocardial infarction, stent thrombosis, and heart failure hospitalization in experimental arm vs. control group.
* Major and minor bleeding in experimental arm vs. control group
* Discontinuation of the drug due to side effects in experimental arm vs. control group A clinical events committee whose members are unaware of study-group assignments will independently adjudicate all potential endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Presenting with acute anterior STEMI
* Severe LV dysfunction (EF<35%) with antero-apical akinesis, dyskinesis, or aneurysm
* WIHTOUT evidence of LV thrombus.

Exclusion Criteria:

* Patients with previous anterior myocardial infarction or LAD revascularization procedures
* Patients with cardiogenic shock
* Patients with LV thrombus
* Patients with advanced CKD (Cr > 2 and those on hemodialysis)
* Recent ICH or major bleed requiring transfusion, low platelet counts <100,000
* History of recent CVA ( within past three months)
* Patients with atrial fibrillation or other indications for chronic anticoagulation
* Pregnant patients and those with hematological disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of LV thrombus formation in the treatment arm vs. control group | one month
  Incidence of LV thrombus formation in the treatment arm vs. control group at 4 week follow up echocardiography. This constitutes the primary endpoint of the trial

SECONDARY OUTCOMES:
Secondary Outcomes | one month
  * composite of death, recurrent myocardial infarction, stent thrombosis, and heart failure hospitalization in the treatment arm vs. control group
  * Major and minor bleeding in the treatment arm vs. control group 3) Discontinuation of the drug due to side effects

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Hakeem Professor of Cardiology, Director Cardiac Catheterization Labs, MD FACC FSCAI FASE, Principal Investigator — NICVD
Locations (1):
- NICVD Pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
We plan on sharing IPD

REFERENCES:
- [Background] Zhang Z, Si D, Zhang Q, Jin L, Zheng H, Qu M, Yu M, Jiang Z, Li D, Li S, Yang P, He Y, Zhang W. Prophylactic Rivaroxaban Therapy for Left Ventricular Thrombus After Anterior ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2022 Apr 25;15(8):861-872. doi: 10.1016/j.jcin.2022.01.285. Epub 2022 Mar 30. PMID 35367170
- [Background] Camaj A, Fuster V, Giustino G, Bienstock SW, Sternheim D, Mehran R, Dangas GD, Kini A, Sharma SK, Halperin J, Dweck MR, Goldman ME. Left Ventricular Thrombus Following Acute Myocardial Infarction: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Mar 15;79(10):1010-1022. doi: 10.1016/j.jacc.2022.01.011. PMID 35272796
- [Background] Bulluck H, Chan MHH, Paradies V, Yellon RL, Ho HH, Chan MY, Chin CWL, Tan JW, Hausenloy DJ. Incidence and predictors of left ventricular thrombus by cardiovascular magnetic resonance in acute ST-segment elevation myocardial infarction treated by primary percutaneous coronary intervention: a meta-analysis. J Cardiovasc Magn Reson. 2018 Nov 8;20(1):72. doi: 10.1186/s12968-018-0494-3. PMID 30404623